CLINICAL TRIAL: NCT01973205
Title: A Multi-center, Randomized, Double-blind, Parallel-group, Single-dose, Placebo-controlled Study Comparing the Efficacy and Safety of a Combination of Acetaminophen and Aspirin vs Placebo in the Acute Treatment of Migraine
Brief Title: Efficacy and Safety of Acetaminophen and Aspirin Versus Placebo in the Acute Treatment of Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 863-P-303
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Acute Migraine
Keywords: Migraine; acetaminophen; aspirin
MeSH Terms: conditions — Migraine Disorders | interventions — Acetaminophen; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 2 placebo tablets matching acetaminophen 250 mg and aspirin 250 mg tablets
  Interventions: Drug: Placebo
- Acetaminophen 250 mg and aspirin 250 mg (Experimental): 2 tablets each containing Acetaminophen 250 mg and aspirin 250 mg
  Interventions: Drug: Acetaminophen 250 mg and Aspirin 250 mg

INTERVENTIONS:
Drug: Acetaminophen 250 mg and Aspirin 250 mg — 2 tablets each containing Acetaminophen 250 mg and Aspirin 250 mg
  Arms: Acetaminophen 250 mg and aspirin 250 mg
Drug: Placebo — 2 placebo tablets matching acetaminophen 250 mg and aspirin 250 mg tablets
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of acetaminophen and aspirin versus placebo in the acute treatment of migraine

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged 18 years and over.
2. International Headache Society (IHS) diagnosis of migraine without aura or typical aura with migraine headache.
3. History of experiencing at least 1, but not more than 8, acute migraine attacks monthly during the previous year.
4. History of at least moderate migraine pain intensity, if left untreated.
5. History of frequently or always experiencing nausea with the migraine attack.

Exclusion criteria:

Subjects eligible for inclusion in this study must not fulfill any of the following criteria:

1. Headache symptoms which may be due to or aggravated by:

   * Recent (within 6 months) head or neck trauma (e.g., whiplash)
   * Head or neck pain secondary to an orthopedic abnormality
   * Cluster headache
   * Specific migraine variants (e.g., basilar-type artery migraine, opthalmoplegic migraine, hemiplegic migraine, migraine aura without headache)
   * Other serious, non-migraine causes of headache (e.g., increased intracranial pressure, intracranial bleeding, meningitis, malignancy)
   * Non-serious, non-migraine causes of headache (e.g., cold, flu, hangover)
2. History of vomiting during more than 20% of migraine attacks.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Lead, Study Director — Novartis Consumer Health
Locations (19):
- United States (19):
  - Birmingham, Alabama
  - Anaheim, California
  - San Francisco, California
  - Fort Lauderdale, Florida
  - Jupiter, Florida
  - Oviedo, Florida
  - West Palm Beach, Florida
  - Evansville, Indiana
  - Ann Arbor, Michigan
  - Berlin, New Jersey
  - Rochester, New York
  - The Bronx, New York
  - Williamsville, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Mt. Pleasant, South Carolina
  - Salt Lake City, Utah
  - Kenosha, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Acetaminophen 250 mg and Aspirin 250 mg
Started | 453 | 447
Completed | 423 | 425
Not Completed | 30 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Acetaminophen 250 mg and Aspirin 250 mg | Total
Number analyzed (Participants) | 453 | 447 | 900
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (12.4) | 39.7 (12.8) | 40.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 351 | 350 | 701
  Male | 102 | 97 | 199
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 48 | 96
  Not Hispanic or Latino | 405 | 399 | 804
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 96 | 105 | 201
  White | 337 | 318 | 655
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 18 | 31
Region of Enrollment [Number; unit: participants]
  United States | 453 | 447 | 900

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Are Pain Free at the 2-hour Assessment
Description: Number of subjects who are pain free at the 2-hour assessment
Time Frame: 2 hours
Population: Number of participants analyzed includes only subjects who treated a migraine (AA: N=408, Placebo: N = 415) and had a non-missing pain free status at 2 hours (AA: N=408, Placebo: N = 415).
Measure: Number; unit: participants
Arm/Group | Placebo | Acetaminophen 250 mg and Aspirin 250 mg
Number analyzed (Participants) | 415 | 408
participants | 69 | 90

2. Primary Outcome: Number of Subjects Who Are Nausea Free at the 2-hour Assessment
Description: Number of subjects who are nausea free at the 2-hour assessment
Time Frame: 2 hours
Population: Number of participants analyzed includes only subjects who treated a migraine (AA: N=408, Placebo: N=415) and had a non-missing nausea free status at 2 hours (AA: N=403, Placebo N= 411).
Measure: Number; unit: participants
Arm/Group | Placebo | Acetaminophen 250 mg and Aspirin 250 mg
Number analyzed (Participants) | 411 | 403
participants | 208 | 244

3. Secondary Outcome: Number of Subjects Who Are Free of Photophobia at the 2-hour Assessment.
Description: Number of subjects who are free of photophobia at the 2-hour assessment.
Time Frame: 2 hours
Population: Number of participants analyzed includes only subjects who treated a migraine (AA: N=408, Placebo: N = 415) and had a non-missing photophobia free status at 2 hours (AA: N=403, Placebo: N = 411).
Measure: Number; unit: participants
Arm/Group | Placebo | Acetaminophen 250 mg and Aspirin 250 mg
Number analyzed (Participants) | 411 | 403
participants | 116 | 127

4. Secondary Outcome: Number of Subjects Who Are Free of Phonophobia at the 2-hour Assessment.
Description: Number of subjects who are free of phonophobia at the 2-hour assessment.
Time Frame: 2 hours
Population: Number of participants analyzed includes only subjects who treated a migraine (AA: N=408, Placebo: N = 415) and had a non-missing phonophobia free status at 2 hours (AA: N=403, Placebo: N = 411).
Measure: Number; unit: participants
Arm/Group | Placebo | Acetaminophen 250 mg and Aspirin 250 mg
Number analyzed (Participants) | 411 | 403
participants | 142 | 164

ADVERSE EVENTS:
Description: Number of participants analyzed includes only subjects who treated a migraine (AA: N=408, Placebo: N = 415)
Arm/Group | Placebo | Acetaminophen 250 mg and Aspirin 250 mg
Serious Adverse Events (participants affected / at risk) | 0/415 | 1/408
Other Adverse Events (participants affected / at risk) | 0/415 | 0/408
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=415) | Acetaminophen 250 mg and Aspirin 250 mg (N=408)
intraductal profilerative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor shall review results communications prior to public release to evaluate the manuscript for accuracy, ascertain whether information (other than the results of the Clinical Trial) is being improperly disclosed, provided information which may have not have yet been made available by the Sponsor, provide input for consideration regarding the content and/or conclusion(s) of the manuscript and determine whether the manuscript discloses any potentially patentable invention(s).